CLINICAL TRIAL: NCT01171404
Title: Long-term Follow-up of Antithrombotic Management Patterns in Acute Coronary Syndrome Patients
Brief Title: Study Evaluating How Patients With Acute Coronary Syndrome Are Managed During 2 Years After Discharge
Acronym: EPICOR
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CEU-DUM-2009/1
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: ACS; Acute Coronary Syndrome; Myocardial Infarction; Unstable Angina; Coronary Artery Disease
Keywords: Acute coronary syndrome; heart attack; myocardial infarction; ACS long-tem follow up; antithrombotic management; quality of life; Antithrombotic
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Angina, Unstable; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients, older than 18, hospitalized within 24 hours of onset of symptoms and diagnosed with UA, STEMI or NSTEMI

SUMMARY:
The aim of this international study is to describe the short- and long-term (i.e. up to 2 years following the index event) antithrombotic management patterns (AMPs) in patients hospitalized for acute coronary syndromes (ST segment elevation myocardial infarction (STEMI), Non-ST-Segment Elevation Acute Coronary Syndrome (NSTE-ACS)), and to document the impact of AMPs in clinical outcomes, economic variables and quality of life in a 'real-life' setting and to compare these between sites, countries and regions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myocardial infarction or unstable angina
* Hospitalized for the first time within 24 hours of onset of symptoms

Exclusion Criteria:

* Presence of any condition/circumstance which in the opinion of the investigator could significantly limit the complete follow up of the patient (e.g. tourist, non-native speaker or does not understand the local language, psychiatric disturbances)
* Current participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized within 24 hours of onset of symptoms and diagnosed with unstable angina (UA), STEMI or non-STEMI(NSTEMI). Patients will be invited to participate by the hospital (Academic or Community) which is going to discharge the patient.
  Participating investigators will belong to hospitals (Academic, Community, with/without cathlab, etc), in the proportion representing the reality of where this kind of patients are managed in each country.
Sampling Method: Probability Sample
Enrollment: 10568 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes (ischemic and bleeding) incidence and time to these clinical outcomes | Longitudinal during 2 years after index event (phone calls to the patients at 6 weeks and each 3 months after index event)

SECONDARY OUTCOMES:
Antithrombotic treatments | Longitudinal during 2 years after index event (phone calls to the patients at 6 weeks and each 3 months after index event)
Use of health care resources | Longitudinal during 2 years after index event (phone calls to the patients at 6 weeks and each 3 months after index event)
Quality of life | At index event (baseline) and then at 6 weeks and each 3 months after index event

CONTACTS AND LOCATIONS:
Overall Officials: Mónica Tafalla, Study Director — Medical Department.AstraZeneca Spain
Locations (410):
- Argentina (16):
  - Research Site, Avellaneda
  - Research Site, Bahía Blanca
  - Research Site, Buenos Aires
  - Research Site, Ciudadela
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, General Roca
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Monteros
  - Research Site, Quilmes
  - Research Site, Rosario
  - Research Site, Salta
  - Research Site, San Isidro
  - Research Site, San Miguel de Tucumán
  - Research Site, San Salvador de Jujuy
- Belgium (32):
  - Research Site, (Jette) Bruxelles
  - Research Site, Aalst
  - Research Site, Antwerp
  - Research Site, Brasschaat
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Chênée
  - Research Site, Dendermonde
  - Research Site, Edegem
  - Research Site, Eeklo
  - Research Site, Genk
  - Research Site, La Louvière
  - Research Site, Leuven
  - Research Site, Lier
  - Research Site, Merksem
  - Research Site, Mol
  - Research Site, Mons
  - Research Site, Montigny-le-Tilleul
  - Research Site, Namur
  - Research Site, Ostend
  - Research Site, Ottignies
  - Research Site, Overpelt
  - Research Site, Roeselare
  - Research Site, Ronse
  - Research Site, Seraing
  - Research Site, Sint-Niklaas
  - Research Site, Soignies
  - Research Site, Tienen
  - Research Site, Tournai
  - Research Site, Turnhout
  - Research Site, Veurne
- Brazil (15):
  - Research Site, Aracaju
  - Research Site, Belo Horizonte
  - Research Site, Blumenau
  - Research Site, Brasília
  - Research Site, Campina Grande do Sul
  - Research Site, Campo Grande
  - Research Site, Curitiba
  - Research Site, Marília
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
  - Research Site, Tatu
  - Research Site, Uberlândia
  - Research Site, Votuporanga
- Denmark (16):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Arhus N
  - Research Site, Esbjerg
  - Research Site, Fredericia
  - Research Site, Frederiksberg
  - Research Site, Haderslev
  - Research Site, Hellerup
  - Research Site, Herning
  - Research Site, Hjørring
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, København Ø
  - Research Site, Odense C
  - Research Site, Silkeborg
  - Research Site, Varde
- Finland (9):
  - Research Site, Espoo
  - Research Site, Helsinki
  - Research Site, Jyväskylä
  - Research Site, Kuopio
  - Research Site, Lahti
  - Research Site, Rovaniemi
  - Research Site, Seinäjoki
  - Research Site, Tampere
  - Research Site, Turku
- France (39):
  - Research Site, Antony
  - Research Site, Argenteuil
  - Research Site, Avignon
  - Research Site, Belfort
  - Research Site, Boulogne-Billancourt
  - Research Site, Bourges
  - Research Site, Brest
  - Research Site, Brive-la-Gaillarde
  - Research Site, Caen
  - Research Site, Chambéry
  - Research Site, Chambray-lès-Tours
  - Research Site, Colmar
  - Research Site, Dijon
  - Research Site, Dunkirk
  - Research Site, Haguenau
  - Research Site, Hopital Civil (strasbourg Cedex)
  - Research Site, La Rochelle
  - Research Site, La Source
  - Research Site, Lagny-sur-Marne
  - Research Site, Le Chesnay
  - Research Site, Le Coudray
  - Research Site, Le Plessis-Robinson
  - Research Site, Marignane
  - Research Site, Marseille
  - Research Site, Metz
  - Research Site, Montfermeil
  - Research Site, Montreuil
  - Research Site, Mulhouse
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Perpignan
  - Research Site, Quimper
  - Research Site, Reims
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Michel-sur-Orge
  - Research Site, Strasbourg
  - Research Site, Suresnes
  - Research Site, Valence
  - Research Site, Vandœuvre-lès-Nancy
- Germany (29):
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Borken
  - Research Site, Cloppenburg
  - Research Site, Coburg
  - Research Site, Detmold
  - Research Site, Dortmund
  - Research Site, Essen
  - Research Site, Esslingen am Neckar
  - Research Site, Greifswald
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Herrsching am Ammersee
  - Research Site, Landshut
  - Research Site, Leverkusen
  - Research Site, Ludwigshafen
  - Research Site, Lübeck
  - Research Site, Mainz
  - Research Site, Merseburg
  - Research Site, Mönchengladbach
  - Research Site, Mühlheim
  - Research Site, Olsberg
  - Research Site, Regensburg
  - Research Site, Rostock
  - Research Site, Stuttgart
  - Research Site, Suhl
  - Research Site, Warendorf
- Greece (12):
  - Research Site, Athens
  - Research Site, Attiki
  - Research Site, Chalcis
  - Research Site, Chania
  - Research Site, Chios
  - Research Site, Edessa
  - Research Site, Elefsina
  - Research Site, Heraklion
  - Research Site, Ioannina
  - Research Site, Larissa
  - Research Site, Pátrai
  - Research Site, Ptolemaida
- Italy (24):
  - Research Site, Ancona
  - Research Site, Catania
  - Research Site, Catanzaro
  - Research Site, Ferrara
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Massa
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Napoli Caserta
  - Research Site, Nuoro
  - Research Site, Ospedale Di Macerata
  - Research Site, Pescara
  - Research Site, Prato
  - Research Site, Rho
  - Research Site, Rimini
  - Research Site, Roma
  - Research Site, Rovigo
  - Research Site, Sassari
  - Research Site, Syracuse
  - Research Site, Treviso
  - Research Site, Udine
  - Research Site, Varese
  - Research Site, Versilia
- Research Site, Luxembourg, Luxembourg
- Mexico (25):
  - Research Site, Cardenas, Tabasco
  - Research Site, Chihuahua City
  - Research Site, Chihuahua, Chihuahua
  - Research Site, Durango
  - Research Site, Durango, Durango
  - Research Site, Guadalajara
  - Research Site, Guadalajara, Jalisco
  - Research Site, Guanajuato City
  - Research Site, León
  - Research Site, Merida, Yucatan
  - Research Site, Mexicali, Baja California
  - Research Site, Mexico City
  - Research Site, Monterrey, Nuevo Leon
  - Research Site, Oaxaca, Oaxaca
  - Research Site, Puebla, Puebla
  - Research Site, Querétaro
  - Research Site, Saltillo Coahuila
  - Research Site, San Luis Potosí City
  - Research Site, Sinaloa, Culiacan
  - Research Site, Tabasco
  - Research Site, Tijuana B.C.
  - Research Site, Toluca, Estado de Mexico
  - Research Site, Torreon Coahuila
  - Research Site, Torreón
  - Research Site, Xalapa, Veracruz
- Netherlands (18):
  - Research Site, Amstelveen
  - Research Site, Amsterdam
  - Research Site, Bergen op Zoom
  - Research Site, Beverwijk
  - Research Site, Delft
  - Research Site, Den Bosh
  - Research Site, Doetinchem
  - Research Site, Goes
  - Research Site, Haarlem
  - Research Site, Heerlen
  - Research Site, Hoofddorp
  - Research Site, Hoogeveen
  - Research Site, Meppel
  - Research Site, Purmerend
  - Research Site, Stadskanaal
  - Research Site, The Hague
  - Research Site, Winterswijk
  - Research Site, Zwolle
- Norway (25):
  - Research Site, Bergen
  - Research Site, Bodø
  - Research Site, Elverum
  - Research Site, Flekkefjord
  - Research Site, Førde
  - Research Site, Gjøvik
  - Research Site, Hamar
  - Research Site, Hammerfest
  - Research Site, Harstad
  - Research Site, Haugesund
  - Research Site, Hønefoss
  - Research Site, Kongsvinger
  - Research Site, Kristiansund N
  - Research Site, Levanger
  - Research Site, Lillehammer
  - Research Site, Lorenskog
  - Research Site, Molde
  - Research Site, Oslo
  - Research Site, Rjukan
  - Research Site, Rud
  - Research Site, Skien
  - Research Site, Tromsø
  - Research Site, Trondheim
  - Research Site, Tynset
  - Research Site, Tønsberg
- Poland (22):
  - Research Site, Bydgoszcz
  - Research Site, Elblag
  - Research Site, Jelenia Góra
  - Research Site, Kalisz
  - Research Site, Koszalin
  - Research Site, Krakow
  - Research Site, Olsztyn
  - Research Site, Opole
  - Research Site, Ostrow Maz.
  - Research Site, Oława
  - Research Site, Poznan
  - Research Site, Pruszków
  - Research Site, Radom
  - Research Site, Sandomierz
  - Research Site, Starogard Gdański
  - Research Site, Słupsk
  - Research Site, Tarnów
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wałbrzych
  - Research Site, Wroclaw
  - Research Site, Włocławek
- Romania (29):
  - Research Site, Alba Iulia
  - Research Site, Arad
  - Research Site, Bacau
  - Research Site, Baia Mare
  - Research Site, Bistriţa
  - Research Site, Brasov
  - Research Site, Brăila
  - Research Site, Bucharest
  - Research Site, Buzău
  - Research Site, Cluj-Napoca
  - Research Site, Constanța
  - Research Site, Craiova
  - Research Site, Drobeta-Turnu Severin
  - Research Site, Focşani
  - Research Site, Galati
  - Research Site, Hunedoara
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Piatra Neamţ
  - Research Site, Piteşti
  - Research Site, Ploieşti
  - Research Site, Râmnicu Vâlcea
  - Research Site, Sibiu
  - Research Site, Slatina
  - Research Site, Suceava
  - Research Site, Târgovişte
  - Research Site, Târgu Mureş
  - Research Site, Timișoara
  - Research Site, Zalău
- Slovenia (2):
  - Research Site, Ljubljana
  - Research Site, Maribor
- Spain (41):
  - Research Site, Alcalá de Henares
  - Research Site, Alcoy
  - Research Site, Alicante
  - Research Site, Aranjuez
  - Research Site, Ávila
  - Research Site, Barcelona
  - Research Site, Baza
  - Research Site, Ciudad Real
  - Research Site, Coslada
  - Research Site, Elche
  - Research Site, Elda
  - Research Site, Ferrol
  - Research Site, Fuenlabrada
  - Research Site, Gandia
  - Research Site, Girona
  - Research Site, Huelva
  - Research Site, Huercal Overa
  - Research Site, Huesca
  - Research Site, Igualada
  - Research Site, León
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Palencia
  - Research Site, Pozoblanco
  - Research Site, Puertollano
  - Research Site, Salamanca
  - Research Site, San Juan
  - Research Site, San Sebastián de los Reyes
  - Research Site, Santiago de Compostela
  - Research Site, Segovia
  - Research Site, Seville
  - Research Site, Tarragona
  - Research Site, Terrassa
  - Research Site, Toledo
  - Research Site, Torrevieja
  - Research Site, Tortosa
  - Research Site, Valencia
  - Research Site, Vélez-Málaga
  - Research Site, Vic
  - Research Site, Villajoyosa
  - Research Site, Zaragoza
- Turkey (Türkiye) (19):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Çanakkale
  - Research Site, Diyarbak?r
  - Research Site, Elaz?g
  - Research Site, Erzurum
  - Research Site, Eskişehir
  - Research Site, Gaziantep
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kayseri
  - Research Site, Konya
  - Research Site, Malatya
  - Research Site, Manisa
  - Research Site, Mersin
  - Research Site, Samsun
  - Research Site, Sivas
  - Research Site, Trabzon
- United Kingdom (29):
  - Research Site, Airdrie
  - Research Site, Antrim
  - Research Site, Basingstoke
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Blackburn
  - Research Site, Blackpool
  - Research Site, Craigavon
  - Research Site, Croydon
  - Research Site, East Kilbride
  - Research Site, Essex
  - Research Site, Glasgow
  - Research Site, Harrow
  - Research Site, Hastings
  - Research Site, Hertfordshire
  - Research Site, High Wycombe
  - Research Site, Kirkcaldy
  - Research Site, Livingston
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Middlesbrough
  - Research Site, Morriston Hospital (Swansea)
  - Research Site, Newcastle upon Tyne
  - Research Site, Peterborough
  - Research Site, Rotherham
  - Research Site, Sheffield
  - Research Site, Stevenage
  - Research Site, Sutton Coldfield
  - Research Site, Worcester
- Venezuela (7):
  - Research Site, Barquisimeto
  - Research Site, Caracas
  - Research Site, Coro
  - Research Site, Maracaibo
  - Research Site, Maracay
  - Research Site, Oriente
  - Research Site, Valencia

REFERENCES:
- [Derived] Huo Y, Van de Werf F, Han Y, Rossello X, Pocock SJ, Chin CT, Lee SW, Li Y, Jiang J, Vega AM, Medina J, Bueno H. Long-Term Antithrombotic Therapy and Clinical Outcomes in Patients with Acute Coronary Syndrome and Renal Impairment: Insights from EPICOR and EPICOR Asia. Am J Cardiovasc Drugs. 2021 Jul;21(4):471-482. doi: 10.1007/s40256-020-00447-5. Epub 2021 Feb 4. PMID 33537947
- [Derived] Martin-Asenjo R, Gregson J, Rossello X, Van de Werf F, Medina J, Danchin N, Pocock S, Bueno H. Number of Antithrombotic Drugs Used Early and In-hospital Outcomes in Acute Coronary Syndromes. J Cardiovasc Transl Res. 2021 Aug;14(4):790-798. doi: 10.1007/s12265-020-10094-5. Epub 2021 Jan 8. PMID 33420682
- [Derived] Stepinska J, Wojtkowska I, Annemans L, Danchin N, Pocock SJ, de Werf FV, Medina J, Bueno H. Long-Term Outcome of Acute Coronary Syndromes in Patients on Chronic Oral Anticoagulants: Data from the EPICOR Study. Curr Vasc Pharmacol. 2020;18(1):92-99. doi: 10.2174/1570161117666181227122355. PMID 30588886
- [Derived] Bardaji A, Leal M, Arrarte V, Garcia-Moll X, Perez de Isla L, Bueno H. Extended dual antiplatelet therapy after acute coronary syndrome in Spain: Results from the EPICOR study. Cardiovasc Ther. 2017 Apr;35(2). doi: 10.1111/1755-5922.12237. PMID 27885830
- [Derived] Bueno H, Pocock S, Danchin N, Annemans L, Gregson J, Medina J, Van de Werf F. International patterns of dual antiplatelet therapy duration after acute coronary syndromes. Heart. 2017 Jan 15;103(2):132-138. doi: 10.1136/heartjnl-2016-309509. Epub 2016 Aug 8. PMID 27504002
- [Derived] Annemans L, Danchin N, Van de Werf F, Pocock S, Licour M, Medina J, Bueno H. Prehospital and in-hospital use of healthcare resources in patients surviving acute coronary syndromes: an analysis of the EPICOR registry. Open Heart. 2016 Feb 24;3(1):e000347. doi: 10.1136/openhrt-2015-000347. eCollection 2016. PMID 27127635
- [Derived] Beauloye C, Vrolix M, Claeys MJ, van de Borne P, Vandendriessche E, Van De Werf F. Pre-hospital management of acute coronary syndrome patients in Belgium and Luxembourg and other Western European countries. Acta Cardiol. 2016 Feb;71(1):15-24. doi: 10.2143/AC.71.1.3132093. PMID 26853249
- [Derived] Zeymer U, Heuer H, Schwimmbeck P, Genth-Zotz S, Wolff K, Nienaber CA; EPICOR Investigators. Guideline-adherent therapy in patients with acute coronary syndromes. The EPICOR registry in Germany. Herz. 2015 Mar;40 Suppl 1:27-35. doi: 10.1007/s00059-014-4161-7. Epub 2014 Nov 7. PMID 25374386
- [Derived] Pocock S, Bueno H, Licour M, Medina J, Zhang L, Annemans L, Danchin N, Huo Y, Van de Werf F. Predictors of one-year mortality at hospital discharge after acute coronary syndromes: A new risk score from the EPICOR (long-tErm follow uP of antithrombotic management patterns In acute CORonary syndrome patients) study. Eur Heart J Acute Cardiovasc Care. 2015 Dec;4(6):509-17. doi: 10.1177/2048872614554198. Epub 2014 Oct 9. PMID 25301783
- [Derived] Bueno H, Danchin N, Tafalla M, Bernaud C, Annemans L, Van de Werf F. EPICOR (long-tErm follow-up of antithrombotic management Patterns In acute CORonary syndrome patients) study: rationale, design, and baseline characteristics. Am Heart J. 2013 Jan;165(1):8-14. doi: 10.1016/j.ahj.2012.10.018. Epub 2012 Nov 20. PMID 23237128